CLINICAL TRIAL: NCT00247000
Title: A Strategy of Home Telehealth for Management of Congestive Heart Failure: STARTEL
Brief Title: A Strategy of Home Telehealth for Management of Congestive Heart Failure(STARTEL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Atlantic Health Sciences Corporation (Other); Heart and Stroke Foundation of Canada (Other); Canada Health Infoway (Other); Continuing Care Nova Scotia (Unknown); Nova Scotia Telehealth Program (Unknown); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDHA005
Record Dates: First submitted 2005-10-30; First posted 2005-11-01 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2006-02

CONDITIONS: Heart Failure
Keywords: Cardiovascular Diseases; Heart Disease; Heart Failure,Congestive; Health Outcomes; Disease Management; Telehomecare; Home Telehealth
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Home teleheatlh for heart failure management
  Interventions: Device: Routine Care in a HF clinic vs Home Telehealth Care for HF
- 2 (Active Comparator): Usual care for the management of Heart Failure
  Interventions: Device: Routine Care in a HF clinic vs Home Telehealth Care for HF

INTERVENTIONS:
Device: Routine Care in a HF clinic vs Home Telehealth Care for HF

SUMMARY:
To demonstrate the safety, feasibility, quality of life, primary caregiver satisfaction, and cost effectiveness of integrated Home Telehealth care versus standard care in a heart failure clinic.

DETAILED DESCRIPTION:
We plan to implement and evaluate a Home Telehealth Care Management System designed to enhance clinical care for congestive heart failure patients who have difficulty with access to care. Unique in this model is that in addition to use of protocol driven interventions (evidence based), the primary care physician is intimately involved in follwo up of patients- with consequent reduction in the fracture of care seen in with attendance in multiple specialty clinics.

In this project, we will evaluate the delivery of care to heart failure patients in Nova Scotia and New Brunswick, with our intervention and the current standard of care, which is the heart failure clinic. Home Telehealth technology will allow patients to be contacted and regularly evaluated in a comprehensive way in their own home, and without the need for a clinic visit. While the Project Team (experienced in heart failure management) will monitor all data, the Family Physician will have first hand access to and right of first treatment when alterations in therapy are needed. This process will be facilitated by the use of protocol driven medical therapy, and delegated medical functions, as well as set-piece education. We hope, with this technology and care plan, to offer the benefits of disease management to this vulnerable patient population while at the same time firmly placing the Family Physician in their central role within the health care system. This program will enable a specific assessment of all aspects of the program, including outcomes, quality of life, professional satisfaction and cost.

ELIGIBILITY:
Patient Population Inclusion Criteria: Patients are eligible for participating in STARTEL if they satisfy all of the following inclusion criteria.

1. Male or female subject's ≥ 18 years of age with a diagnosis of Heart Failure
2. Subject must reside in either the Province of Nova Scotia or New Brunswick
3. Subject has been hospitalized for heart failure during the past two years or has a known history of heart failure for a minimum of two years.
4. Subject must have a dedicated working telephone line in their primary place of residence.
5. Subject must have a grounded electrical power supply in their primary place of residence.
6. Primary care physician provides their agreement to participate in STARTEL

Exclusion Criteria: Patients are not eligible for participating in STARTEL if they meet any of the following exclusion criteria.

1. Inability to understand the English or French language or understand the study and provide informed consent.
2. Absence of a suitable area to conduct the home telehealth visit in the patient's place of residence.
3. Physical impairment, which would prohibit the successful completion of a home telehealth visit, including attachment of the peripheral equipment (BP cuff, ability to stand on a scale, etc).
4. In cases 1 & 3 only: a live in caregiver whose presence may overcome these limitations may allow the patient to be included in the study, however, only the patient's next of kin or duly appointed guardian (with documentation and with patient assent) may provide informed consent to participate).
5. Subject has a planned cardiac procedure such as open-heart surgery or percutaneous coronary intervention (PCI) within the next 6 months.
6. Subject has had cardiac surgery, percutaneous coronary intervention or a diagnosis of acute myocardial infarction within 1 month before randomization).
7. Condition where existing routine follow up occurs more than once weekly (i.e. hemodialysis, cancer treatment including: chemotherapy/radiation treatment). .
8. Patient is institutionalized (includes chronic care facility)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-11; Primary Completion 2009-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
A composite of total all-cause hospitalizations and total mortality at one year. | 1 year

SECONDARY OUTCOMES:
Heart failure morbidity and mortality | 1 year
Cardiovascular hospitalization | 1 year
Total number days in hospital | 1 year
Total outpatient physician visits | 1 year
Number of non-scheduled health visits outside the home | 1 year
Total inpatient and outpatient health care costs | 1 year
Kansas City Cardiomyopathy Quality of Life Score | 1 year
Total medication related costs | 1 year
Medication adherence(by prescription filling data) | 1 year
Patient satisfaction as measured on Likert scale(1-10) | 1 year
Primary care physician satisfaction (Likert scale) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan G Howlett, M.D.,FRCPC, Principal Investigator — Capital District Health Authority, QEII Health Sciences Centre
Locations (1):
- New Brunswick Heart Centre, Atlantic Health Sciences Corporation, Saint John, New Brunswick, Canada